CLINICAL TRIAL: NCT07286123
Title: Gender Affirming Vaginoplasty With Tubularized Augmented Peritoneal Cap (TAPCap) Utilizing Fish Skin Xenograft (Kerecis™)
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kerecis Ltd. (Industry)
Responsible Party: Principal Investigator, Shubham Gupta, Professor, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20250076
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gender Dysphoria, Adult
Keywords: xenograft; gender affirming vaginoplasty; bottom surgery
MeSH Terms: conditions — Gender Dysphoria | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals receiving vaginoplasty: Individuals requiring graft-based vaginoplasty
  Interventions: Procedure: Tubularized augmented peritoneal cap vaginoplasty; Procedure: Biopsy

INTERVENTIONS:
Procedure: Tubularized augmented peritoneal cap vaginoplasty — In this surgery, the distal portion of the neovagina is constructed using inverted penile skin, the proximal portion is made of peritoneal tissue. The area in between peritoneal tissue and penile skin is lined with the Kerecis graft in this standard of care surgery.
Procedure: Biopsy — Biopsies will be obtained at 6 months post-op from the distal, middle, and proximal portions of the neovagina.

SUMMARY:
Bottom gender affirming surgery is one of the key steps towards aligning the physical appearance and gender identity in transgender women. This surgery not only helps in reducing gender dysphoria but also significantly improves the quality of life and psychological well-being of the patients. The basic steps of bottom surgery typically involve the creation of a vagina using the skin from genital organs like the testes and penis, construction of the clitoris and labia. This complex surgery aims to create a functional and aesthetically pleasing vaginal canal that allows for sexual activity, urinary function, and a natural appearance.

As part of routine care, a special graft (skin-like material) called Kerecis™ is used to line the middle part of the vagina. It is made from North Atlantic cod skin that is treated in the laboratory and made suitable for surgery purposes. It can be used instead of skin. This graft has been given permission by the Food and Drug Administration (FDA) for marketing the US.

This study aims to identify changes in healing parameters following Kerecis™ based vaginoplasty. Up to 20 participants for this study.

Participants will be asked to fill out study questionnaires during follow-up visits at post-op week 2, week 12, month , and year 1.

At the 6 month post-op follow up, punch biopsies will be obtained from the deepest part, middle part, and the vaginal part most near to the vaginal opening parts to check the healing process using a microscope. The punch biopsies will be 1/8th inch x 1/8th inch each.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-99
* Transgender women planning for gender affirming robotic vaginoplasty with TAPCap technique

Exclusion Criteria:

* Patients requiring Kerecis for Revision Vaginoplasty
* Surgery candidates having Zero depth vaginoplaty (ZDV)
* Non-Gender Affirming Vaginoplasty
* Cases requiring the utilization of off-the-shelf grafts other than Kerecis
* Allergy to fish products
* Allergy to local anesthetic (1% lidocaine with epinephrine injection)

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are only eligible if assigned sex at birth is male, and diagnosed with gender dysphoria.
Study Population: Individuals requiring graft-based vaginoplasty
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Degree of Neovaginal Epithelialization | Six months post-op
  Degree of epithelialization of each sample biopsy. Biopsies are obtained from the proximal segment (peritoneal portion), middle segment (Xenograft portion), and, distal segment (penile skin portion) of the neovagina.
  Grade 0: No epithelialization Grade 1 : Minimal epithelialization Grade 2: Moderate epithelialization Grade 3: Significant epithelialization
Change in Vaginal Diameter | Post-op week 2, week, 12, month 6, and year 1
  The participants' vaginal diameter is calculated based on the largest tolerated vaginal dilator size (Soul Source; CA, USA) . Measurements are reported in centimeters (cm).
Change in Vaginal Depth | Post-op week 2, week, 12, month 6, and year 1
  The participants' vaginal depth are calculated based on the largest tolerated vaginal dilator (Soul Source, CA, USA). Measurements are reported in centimeters (cm).
Change in quality of life as measured by the Short-Form 36 (SF-36) | Week 2, Week 12, Month 6, and year 1 post-op
  This is a validated questionnaire measuring health-related quality of life through eight domains, covering physical and mental well-being. It's widely used in healthcare to assess overall health perception and functional status. With higher scores indicating greater quality of life.
Change in Pain as measured by the Brief Pain Inventory - Short Form (BPI-SF) | Week 2, Week 12, Month 6, and year 1 post-op
  This is a concise validated questionnaire used to evaluate the severity and impact of pain experienced by individuals. It consists of questions that assess the intensity of pain at its worst, least, average, and current levels, as well as its interference with various aspects of daily life such as general activity, mood, walking ability, work, relationships, and enjoyment of life. Higher scores indicate worse outcomes.
Change in Pain as measured by the The Female Genitourinary Pain Index (GUPI) | Week 2, Week 12, Month 6, and year 1 post-op
  This is a validated questionnaire used to assess symptoms related to genitourinary pain in women. It includes questions covering pain severity, urinary symptoms, and impact on quality of life, providing clinicians with a standardized tool to evaluate and monitor participants' symptoms and treatment responses in these chronic pain conditions. Higher scores indicate worse outcomes.
Change in overall perception of improvement as measured by the PGI-I (Patient Global Impression of Improvement) | Week 2, Week 12, Month 6, and year 1 post-op
  This is a patient-reported scale that measures how individuals perceive their overall improvement after treatment, offering clinicians insight into treatment effectiveness from the participant's viewpoint. Lower scores indicate better outcomes.
Change in sexual function of improvement as measured by the Female Sexual Function Index (FSFI) | Month 6, and year 1 post-op
  This is a validated 19-item questionnaire assessing six domains of female sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. Each domain is scored, and the total score reflects overall sexual function, with higher scores indicating better function. It is used in clinical and research settings to evaluate sexual health and the impact of treatments. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Gupta, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No